CLINICAL TRIAL: NCT02975076
Title: Radix/Rhizoma Notoginseng Extract (Sanchitongtshu) Plus Asprine for Minor Ischemic Stroke or Transient Ischemic Attack: A Randomized Double-blind Placebo-controlled Study
Brief Title: Sanchitongtshu Plus Asprine for Minor Ischemic Stroke or Transient Ischemic Attack: A Randomized Double-blind Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: XH-16-037
Record Dates: First submitted 2016-11-18; First posted 2016-11-29 (Estimated); Last update posted 2016-11-29 (Estimated); Status verified 2016-11

CONDITIONS: Stroke, Acute; Ischemic Attack, Transient
Keywords: Sanchitongshu; Acute Minor Stroke; Transient Ischemic Attack
MeSH Terms: conditions — Stroke; Ischemic Attack, Transient | interventions — Aspirin; Clopidogrel

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sanchitongshu & placebo of lopidogrel (Experimental): sanchitongshu 1 capsule each time ,three times a day and Aspirin 75mg for 90 days ; placebo of clopidogrel 75mg daily for 21 days after randomization
  Interventions: Drug: Sanchitongshu; Drug: Aspirin; Drug: placebo of clopidogrel
- placebo of Sanchitongshu & lopidogrel (Placebo Comparator): placebo of sanchitongshu1 capsule each time ,three times a day and Aspirin 75mg for 90 days;clopidogrel 75mg per day for 21 days after randomization
  Interventions: Drug: placebo of Sanchitongshu; Drug: Aspirin; Drug: Clopidogrel

INTERVENTIONS:
Drug: Sanchitongshu — The study drugs were manufactured according to Good Manufacturing Practice (GMP) by the Pharmaceutical Factory of Chengdu Huasun Group Inc. Ltd. and presented in the form capsules. Every Sanchitongshu capsule weighed 200 mg, contained 100 mg of panaxatriol saponin (PTS) and 100 mg inactive excipient (starch). PTS comprised of dried extracts from roots of Radix Notoginseng, and had been standardised with respect to Ginsenoside Rg1 (50%), Ginsenoside Re (6%), Notoginsenoside R1 (11%). The amounts of the active ingredients were determined by analytical RP-HPLC using an acetonitrile-water gradient system as mobile hase. The peaks were detected by UV-DAD.
  Other Names: Radix/Rhizoma Notoginseng extract
  Arms: Sanchitongshu & placebo of lopidogrel
Drug: placebo of Sanchitongshu — The Sanchitongshu placebo capsule contained dark brown muscovado sugar and the same inactive excipient (starch).
  Arms: placebo of Sanchitongshu & lopidogrel
Drug: Aspirin
  Other Names: Aspirin Enteric-coated Tablets
Drug: Clopidogrel
  Other Names: Clopidogrel Bisulfate
  Arms: placebo of Sanchitongshu & lopidogrel
Drug: placebo of clopidogrel
  Arms: Sanchitongshu & placebo of lopidogrel

SUMMARY:
Agents of sanchi have been widely used as a complementary medicine for stroke in China. Sanchitongshu is a new Chinese patent medicine extracted from sanchi which has stronger anti-platelet activity than other agents of sanchi. The investigators's aim was to investigate the synergistic action of aspirin combined with sanchitongshu capsule in the treatment of patients with minor ischemic stroke and transient ischemic attack.

DETAILED DESCRIPTION:
Transient ischemic attack (TIA) and acute minor ischemic stroke are common and often lead to disabling events. In China, there are approximately 3 million new strokes every year, and approximately 30% of them are minor ischemic strokes. The incidence of TIA in China has not been determined, but on the basis of the incidence in other countries, there are probably more than 2 million TIAs annually in China. The risk of another stroke occurring after a TIA or minor stroke is high, with approximately 10 to 20% of patients having a stroke within 3 months after the index event; most of these strokes occur within the first 2 days. The role of antiplatelet therapy for secondary stroke prevention has been well established.

As yet, aspirin is the only antiplatelet agent that has been studied in the acute phase of stroke, during which its benefit is modest. Clopidogrel in High-Risk Patients with Acute Nondisabling Cerebrovascular Events (CHANCE) trial shows that among patients with high-risk TIA or minor ischemic stroke who are initially seen within 24 hours after symptom onset, treatment with clopidogrel plus aspirin for 21 days, followed by clopidogrel alone for a total of 90 days, is superior to aspirin alone in reducing the risk of subsequent stroke events. The combination of clopidogrel with aspirin did not cause more hemorrhagic events in this patient population than aspirin alone. The analytical results provided basis for the synergistical effect of Aspirin and clopidogrel in inhibiting platelet aggregation. However, long term use of clopidogrel bring people financial burden so that the patients have less compliance of medication. Therefore, the investigators need to explore new treatment for more effective, safe and economic.

Sanchi is one of the most widely used herbal medicine in China for ischemic stroke, of which panax notoginseng saponins (PNS) are the main active components. Previously there were lots of clinical trials on agents of PNS for ischemic stroke in China and had positive results. Sanchitongshu capsule is a new Chinese patent medicine extracted from sanchi. 80% of the ingredients in sanchi-tongshu capsule are panaxatriol saponins (PTS) and 60% of PTS are Rg1 which has strongest anti-platelet activity of all the PNS. PTS were proven by experiment and phase III clinical trials to have antithrombosis effect through mechanisms of inhibiting platelet aggregation, decreasing blood viscosity, strengthening activities of fibrinolysis system, and promoting vascular endothelial NO releasing. More recent experimental studies indicated anti-inflammatory and neuroprotective effect of PTS. Compared with other agents of Sanchi, Sanchitongshu capsule contains higher purity of PTS and Rg1. Thus, Sanchitongshu capsule theoretically should be vigorous in improving ischemic status after ischemic stroke.

Include, the investigators will investigate the synergistic action of aspirin combined with sanchitongshu capsule in the treatment of patients with minor ischemic stroke and transient ischemic attack.

ELIGIBILITY:
Inclusion Criteria:

1. age of 40 years to 80 years
2. diagnosis of an acute minor ischemic stroke or transient ischemic attack; and ability to start the study drug within 24 hours after symptom onset, which was defined as the point at which the patient reported no longer being in a normal condition. Acute minor stroke was defined by a score of 3 or less at the time of randomization on the National Institutes of Health Stroke Scale(NIHSS). TIA was defined as focal brain ischemia with resolution of symptoms within 24 hours after onset plus a moderate-to-high risk of stroke recurrence(defined as a score≥4 at the time of randomization on the ABCD2). All patients were confirmed by brain CT or MRI.
3. Patients had ability to accept the medicine and rules of the research.
4. Patients had no serious complications and had normal renal function and liver function.

Exclusion Criteria:

1. age younger than 40 and older than 80
2. Patients need thrombolysis
3. hemorrhage; other conditions, such as vascular malformation, tumor, abcess, or other major nonischemic brain disease
4. isolated sensory symptoms(e.g., numbness), isolated visual changes, or isolated dizziness or vertigo without evidence of acute infarction on baseline CT or MRI of the head
5. a score of more than 2 on the modified Rankin scale(scores ranges from 0(no symptoms) to 6(death))immediately before the occurrence of the index ischemic stroke or TIA, indicating moderate disability or worse at baseline
6. TIA or minor stroke caused by angiography or surgery
7. a clear indication for anticoagulation therapy(presumed cardiac source of embolus, such as atrial fibrillation or prosthetic cardio valve)
8. anticipated requirement for long-term nonstudy antiplatelet drugs or for non steroidal antiinflammatory drugs affecting platelet function
9. accompanied with severe disorders of heart, liver, and kidney
10. severe noncardiovascular coexisting condition, with a life expectancy of less than 3 months.
11. history of hemorrhage or bleeding tendency of other system( such as thrombocytopenic purpura)
12. gastrointestinal bleeding or major surgery within the previous 3 months
13. planned or probable revascularization(any angioplasty or vascular surgery)within 3 months after.Operation or Interventional Therapy require discontinuation of study drug
14. Aspirin, clopidogrel or notoginseng allergy
15. a history of alcoholism or drug abuse in past 12 months
16. pregnant and lactating women, or women of childbearing age without taking any effective contraceptive measures
17. patients have other serious disease or abnormal laboratory results that is unfavorable to join the research
18. patients receiving other investigational drugs or devices
19. incomprehension of the character and category of the research and unable to follow the research plan

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2016-12; Primary Completion 2019-11 (Estimated); Study Completion 2019-11 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients with the180-day new vascular events, defined as any event of the following: Any stroke (ischemic or hemorrhage) | 180 days

SECONDARY OUTCOMES:
Percentage of patients with the 180-day new clinical vascular events (ischemic stroke/ hemorrhagic stroke/ TIA/ MI/ vascular death) as a cluster and evaluated individually | 180 days
Modified Rankin Scale score changes (continuous) and dichotomized at percentage with score 0-2 vs. 3-6 at 180 days follow-up | 180 days
Further efficacy exploratory analysis:Impairment (changes in NIHSS scores at 180 days follow-up) | 180 days
Further efficacy exploratory analysis:Impairment (changes in Barthel Index at 180 days follow-up) | 180 days
Further efficacy exploratory analysis: stroke impact scale | 180 days
Efficacy endpoint will also be analyzed stratified by etiological subtypes | 180 days
death from any cause | 180 days
Severe bleeding incidence (GUSTO definition), including fatal bleeding and symptomatic intracranial hemorrhage. | 180 days
Incidence symptomatic and asymptomatic intracranial hemorrhagic events at 180 days | 180 days
Incidence Intracranial hemorrhage events at 180 days | 180 days

CONTACTS AND LOCATIONS:
Overall Officials: Xinhua Hospital, Study Director — Xinhua Hospital, Shanghai Jiao Tong University School of Medicine

IPD SHARING:
Plan to Share IPD: Yes